CLINICAL TRIAL: NCT05654090
Title: A Randomized, Single-dose, Two-way Crossover Study to Evaluate Bioequivalence of Two Formulations of Cefoperazone Sodium and Sulbactam Sodium Combination (1/1 g/Vial) After Intravenous Infusion of 1 g Cefoperazone Sodium and 1 g Sulbactam Sodium in Healthy Volunteers Under Fasting Conditions
Brief Title: Evaluate Bioequivalence of Burotam (1/1 g/Vial)
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Yung Shin Pharm. Ind. Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: YSP-RNH3002-01
Record Dates: First submitted 2022-12-08; First posted 2022-12-16 (Actual); Last update posted 2023-02-01 (Actual); Status verified 2022-08

CONDITIONS: Infectious Diseases
MeSH Terms: conditions — Communicable Diseases | interventions — Cefoperazone; Sulbactam

STUDY DESIGN:
Intervention Model Description: An open-label, randomized, balanced, two-treatment, two-period, twosequence, single dose, two-way crossover study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- cefoperazone sodium and sulbactam sodium (Product name:Burotam) (Experimental): Single dose Burotam
  Interventions: Drug: cefoperazone sodium and sulbactam sodium
- cefoperazone sodium and sulbactam sodium (Product name:Brosym) (Active Comparator): Single dose Brosym
  Interventions: Drug: cefoperazone sodium and sulbactam sodium

INTERVENTIONS:
Drug: cefoperazone sodium and sulbactam sodium — Pharmacokinetic study under fasting conditions

SUMMARY:
A randomized, single-dose, two-way crossover study to evaluate bioequivalence of two formulations of cefoperazone sodium and sulbactam sodium combination (1/1 g/vial) after intravenous infusion of 1 g cefoperazone sodium and 1 g sulbactam sodium in healthy volunteers under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adult male or female subjects between 20-45 years of age (inclusive) at the screening visit.
2. Body mass index (BMI) between 18 and 27 kg/m2 (not inclusive) at the screening visit.
3. Acceptable medical history and physical examination including:

   * no particular clinically significant abnormalities in ECG results within six months prior to Period I dosing.
   * no particular clinical significance in general disease history within two months prior to Period I dosing.
4. Acceptable biochemistry determinations (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes AST (SGOT), ALT (SGPT), γ-GT, alkaline phosphatase, total bilirubin, albumin, glucose, BUN, uric acid, creatinine, total cholesterol and triglyceride (TG).
5. Acceptable hematology (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes hemoglobin, hematocrit, red blood cell count, white blood cell count with differentials and platelets.
6. Acceptable urinalysis (within normal limits or considered by the investigator or physician to be of no clinical significance) within two months prior to Period I dosing, which includes pH, blood, glucose, ketones, bilirubin and protein.
7. Female of childbearing potential practicing an acceptable method of birth control for the duration of the study.
8. Have signed the written informed consent to participate in the study.

Exclusion Criteria:

1. A clinically significant disorder involving the cardiovascular, respiratory, hepatic, renal, urinary tract, gastrointestinal, immunologic, hematologic, endocrine or neurologic system(s) or psychiatric disease.
2. A clinically significant illness or surgery within four weeks prior to Period I dosing.
3. History of gastrointestinal obstruction, inflammatory bowel disease, gallbladder disease, pancreas disorder over last two years or history of gastrointestinal tract surgery over last five years.
4. History of kidney disease or urination problem over last two years deemed by the investigator to be clinically significant.
5. Known or suspected history of drug abuse within lifetime.
6. History of alcohol addiction or abuse within last five years or use of more than 7 units of alcohol per week within two weeks prior to dosing. (1 unit of alcohol = 10 g of alcohol or about 350 mL of beer or about 83 mL of red wine or about 30 mL of beverage containing 40% (v/v) alcohol).
7. History of allergic response(s) to palonosetron or any other related drugs.
8. Evidence of chronic or acute infectious diseases.
9. Positive result for serum hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCVAb), or human immunodeficiency virus (HIV).
10. Female subjects demonstrating a positive pregnancy screen prior to the study.
11. Female subjects who are currently breastfeeding.
12. Taking any drug known to induce or inhibit hepatic drug metabolism within four weeks prior to Period I dosing. Examples of inducers include: piperidines, carbamazepine, dexamethasone and rifampin. Examples of inhibitors include: cimetidine, diphenhydramine, fluvastatin, methadone and ranitidine.
13. Taking any prescription medications within four weeks or any nonprescription medications (excluding flu vaccination) within two weeks prior to Period I dosing.
14. Use of any investigational drug within four weeks prior to Period I dosing.
15. Use of any COVID-19 vaccine within seven days prior to Period I dosing.
16. Donating more than 250 mL of blood within two months prior to Period I dosing or donating plasma (e.g. plasmapheresis) within two weeks prior to Period I dosing.
17. Any other medical reason as determined by the investigator.

Ages: 20 Years to 20 Years | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Estimated)
Dates: Start 2022-08-25 (Actual); Primary Completion 2022-11-18 (Actual); Study Completion 2023-02-20 (Estimated)

PRIMARY OUTCOMES:
Peak plasma concentration (Cmax) | 0 (pre-dose), 5, 10 minutes after the start of infusion, immediately after the end of infusion (15 minutes after the start of infusion), and 5, 15, 30, and 45 minutes, and 1.75, 2.75, 3.75, 4.75, 5.75, 7.75, and 11.75 hours after the end of infusion
Area under the concentration-time curve from time zero to time of last quantifiable | 0 (pre-dose), 5, 10 minutes after the start of infusion, immediately after the end of infusion (15 minutes after the start of infusion), and 5, 15, 30, and 45 minutes, and 1.75, 2.75, 3.75, 4.75, 5.75, 7.75, and 11.75 hours after the end of infusion
Area under the concentration-time curve from time zero to infinity (AUC 0-∞) | 0 (pre-dose), 5, 10 minutes after the start of infusion, immediately after the end of infusion (15 minutes after the start of infusion), and 5, 15, 30, and 45 minutes, and 1.75, 2.75, 3.75, 4.75, 5.75, 7.75, and 11.75 hours after the end of infusion

CONTACTS AND LOCATIONS:
Locations (1):
- Taichung Veterans General Hospital, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No